CLINICAL TRIAL: NCT03453125
Title: Improving Learning in Hispanics With TBI or MS: A Pilot Trial
Brief Title: Improving Learning in Hispanics With TBI or MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: Instituto Vocacional Enrique Díaz de León A.C., Guadalajara, Mexico (Unknown)
Responsible Party: Principal Investigator, Denise Krch, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-799-13
Record Dates: First submitted 2018-02-21; First posted 2018-03-05 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: TBI (Traumatic Brain Injury) or MS (Multiple Sclerosis)
Keywords: cognitive rehabilitation; memory
MeSH Terms: conditions — Brain Injuries, Traumatic; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spanish mSMT Experimental Treatment (Experimental): Administered by computer and paper and pencil.
  Interventions: Behavioral: Spanish modified Story Memory Technique (mSMT)
- Spanish mSMT Control Treatment (Active Comparator): Administered by computer and paper and pencil.
  Interventions: Behavioral: Spanish modified Story Memory Technique (mSMT)

INTERVENTIONS:
Behavioral: Spanish modified Story Memory Technique (mSMT)

SUMMARY:
The goal of this study is to establish that a memory retraining protocol, originally developed for English-speakers, and translated into Spanish, is effective.

DETAILED DESCRIPTION:
A pilot study will be conducted to carry out this validation and resolve any methodological concerns in the translated protocol. 20 Spanish-speaking Hispanics at least one year post-traumatic brain injury (TBI) and 20 Spanish-speaking Hispanics with multiple sclerosis (MS), both with an objective deficit in learning and memory will be recruited. Baseline assessment includes neuropsychological evaluation using traditional measures as well as completion of a number of questionnaires designed to measure everyday memory and everyday functioning. Subjects are randomly assigned to either the experimental or control groups. Experimental and control treatments includes two 45-60 minute sessions, twice per week, for 5 weeks. Follow-up assessment includes a neuropsychological evaluation using traditional measures as well as completion of a number of questionnaires designed to measure everyday memory and everyday functioning. Protocol efficacy will be determined by improvements between baseline and follow-up on an objective measure of learning and memory.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 65
* Spanish is my dominant language, and I have had a traumatic brain injury or I have multiple sclerosis.

Exclusion Criteria:

* Participants with major depressive disorder, schizophrenia, bipolar disorder I or II
* MS subjects: Individuals with a history of head injury, stroke, seizures, or any other significant neurological history will not be included in the study.
* TBI subjects: Individuals must have sustained a TBI at least one year prior to enrollment in the study protocol. Individuals with a history of significant neurological insult other than TBI (e.g. premorbid epilepsy, multiple sclerosis, Alzheimer's disease) will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09-25 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Total learning post-treatment (covarying for baseline performance) | 7 weeks (between pre- and post testing)
  Comparison between treatment and control groups on post-treatment Hopkins Verbal Learning Test (HVLT) learning score, covarying for baseline HVLT performance.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chiaravalloti, PhD, Study Director — Kessler Foundation
Locations (2):
- Kessler Foundation, East Hanover, New Jersey, United States
- Hospital Aita Menni, Arrasate / Mondragón, Spain

IPD SHARING:
Plan to Share IPD: Undecided